CLINICAL TRIAL: NCT01220180
Title: Post Marketing Surveillance Study For Observing Safety And Efficacy Of Lyrica
Brief Title: Lyrica (Pregabalin) Korean Post Marketing Surveillance Study
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A0081138
Record Dates: First submitted 2010-10-07; First posted 2010-10-13 (Estimated); Results first posted 2011-12-08 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2011-11

CONDITIONS: Epilepsy; Neuropathic Pain; Fibromyalgia; Post-market Surveillance
Keywords: epilepsy; neuropathic pain; fibromyalgia; post-market surveillance; prospective observational
MeSH Terms: conditions — Epilepsy; Neuralgia; Fibromyalgia | interventions — Pregabalin

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Epilepsy
  Interventions: Drug: pregabalin (Lyrica)
- Neuropathic Pain
  Interventions: Drug: pregabalin (Lyrica)
- Fibromyalgia
  Interventions: Drug: pregabalin (Lyrica)

INTERVENTIONS:
Drug: pregabalin (Lyrica) — Pregabalin treatment can be started with a dose of 150 mg per day. Based on individual subject response and tolerability, the dosage may be increased to 300 mg per day after 1 week. The maximum dosage of 600 mg per day may be achieved after an additional week.
  Groups: Epilepsy
Drug: pregabalin (Lyrica) — Peripheral neuropathic pain: Pregabalin treatment can be started at a dose of 150 mg per day. Based on individual subject response and tolerability, the dosage may be increased to 300 mg per day after an interval of 3 to 7 days, and if needed, to a maximum dose of 600 mg per day after an additional 7-day interval.
  Central neuropathic pain: Pregabalin treatment can be started at a dose of 150 mg per day. Based on individual subject response and tolerability, the dosage may be increased to 300 mg per day after an interval of 1 week, and if needed, to a maximum dose of 600 mg per day after an additional 1 week interval. In case that tolerability could not be shown in the targeted daily dose, dose reduction may be considered.
  Groups: Neuropathic Pain
Drug: pregabalin (Lyrica) — The recommended dose of pregabalin for fibromyalgia is 300 to 450 mg/day. Dosing should begin at 75 mg two times a day (150 mg/day) and may be increased to 150 mg two times a day (300 mg/day) within 1 week based on efficacy and tolerability. Subjects who do not experience sufficient benefit with 300 mg/day may be further increased to 225 mg two times a day (450 mg/day). Treatment with doses above 450 mg/day is not recommended.
  Groups: Fibromyalgia

SUMMARY:
This study collects post-marketing safety and efficacy surveillance data in real world clinical use of pregabalin for its approved indications in Korea.

DETAILED DESCRIPTION:
continuous patients with target disorders in collaborating institutions

ELIGIBILITY:
Inclusion Criteria:

* Any patient treated with pregabalin for an approved indication by Korean Food and Drug Administration

Exclusion Criteria:

* Non-consenting
* Hypersensitivity to the active substance or to any of the excipients
* galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Korean adult patients with epilepsy, neuropathic pain or fibromyalgia, prescribed pregabalin for within label use
Sampling Method: Non-Probability Sample
Enrollment: 4175 (Actual)
Dates: Start 2006-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081138&StudyName=Lyrica%20%28Pregabalin%29%20Korean%20Post%20Marketing%20Surveillance%20Study%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin: Pregabalin capsules administered orally starting with a dose of 150 milligram per day (mg/day) which could be increased up to a maximum dosage of 600 mg/day in adult participants with epilepsy and neuropathic pain (peripheral or central); and the recommended dose for fibromyalgia was 300 to 450 mg/day.
Period: Overall Study
Arm/Group | Pregabalin
Started | 4175
Treated | 4174
Completed | 3968
Not Completed | 207
Not completed — Lost to Follow-up | 76
Not completed — Other | 72
Not completed — Adverse Event | 35
Not completed — Lack of Efficacy | 22
Not completed — Death | 1
Not completed — Randomized but not treated | 1

BASELINE CHARACTERISTICS:
Groups:
- Pregabalin: Epilepsy: Pregabalin capsules administered orally starting with a dose of 150 mg/day which could be increased up to a maximum dosage of 600 mg/day in adult participants with epilepsy.
- Pregabalin: Neuropathic Pain: Pregabalin capsules administered orally starting with a dose of 150 mg/day which could be increased up to a maximum dosage of 600 mg/day in adult participants with Neuropathic pain (NeP).
- Pregabalin: Fibromyalgia: Pregabalin capsules administered orally starting with a dose of 300 to 450 mg/day in adult participants with fibromyalgia.
- Total: Total of all reporting groups
Arm/Group | Pregabalin: Epilepsy | Pregabalin: Neuropathic Pain | Pregabalin: Fibromyalgia | Total
Number analyzed (Participants) | 787 | 3266 | 121 | 4174
Age, Customized [Number; unit: Participants]
  Less than 20 years | 37 | 2 | 0 | 39
  20 to 29 years | 192 | 26 | 3 | 221
  30 to 39 years | 158 | 105 | 8 | 271
  40 to 49 years | 146 | 409 | 30 | 585
  50 to 59 years | 119 | 840 | 36 | 995
  60 to 69 years | 89 | 1094 | 28 | 1211
  Greater than and equal to 70 years | 46 | 790 | 16 | 852
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 364 | 1689 | 83 | 2136
  Male | 423 | 1577 | 38 | 2038

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving 28 Days Seizure Free Period in Intent-to Treat (ITT) Population
Description: Participants were regarded as seizure-free if no seizures (partial or other) were reported for the participant during the period of 28 days in the study.
Time Frame: Baseline through Week 12
Population: ITT population included participants who received at least 1 dose of the study medication and indication of use was epilepsy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Pregabalin: Pregabalin capsules administered orally starting with a dose of 150 mg/day which could be increased up to a maximum dosage of 600 mg/day in adult participants with epilepsy and neuropathic pain (peripheral or central); and the recommended dose for fibromyalgia was 300 to 450 mg/day.
Arm/Group | Pregabalin
Number analyzed (Participants) | 644
Percentage of participants | 66.30 [62.65 to 69.96]

2. Primary Outcome: Percentage of Participants Achieving 28 Days Seizure Free Period in Per Protocol (PP) Population
Description: as for outcome 1
Time Frame: Baseline through Week 12
Population: PP population included participants who received the study medication for at least 12 weeks and indication of use was epilepsy.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 575
Percentage of participants | 67.13 [63.29 to 70.97]

3. Primary Outcome: Percentage of Participants With Improvement in Seizure Frequency in ITT Population
Description: Percentage of participants with improvement in seizure frequency of greater than or equal to 75%; greater than or equal to 50% to 74%; 0% to 49% were considered.
Time Frame: Baseline through Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 644
Percentage of participants
  Greater than or equal to 75% | 55.75
  Greater than or equal to 50% to 74% | 28.57
  0% to 49% | 14.13
  Worsening | 1.55

4. Primary Outcome: Percentage of Participants With Improvement in Seizure Frequency in PP Population
Description: as for outcome 3
Time Frame: Baseline through Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 575
Percentage of participants
  Greater than or equal to 75% | 57.22
  Greater than or equal to 50% to 74% | 29.39
  0% to 49% | 12.52
  Worsening | 0.87

5. Primary Outcome: Change From Baseline in Daily Pain Score for NeP in ITT Population at Week 6
Description: Daily Pain Rating Score (DPRS): participant rated 11-point Likert scale ranging from 0 (no pain) to 10 (worst possible pain) during past 24-hour period. Higher score indicates greater level of pain.
Time Frame: Baseline and Week 6
Population: ITT population included participants who received at least 1 dose of the study medication and indication of use was NeP.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 3210
Units on a scale
  Baseline | 5.61 (1.77)
  Change at Week 6 | -3.02 (1.79)
Statistical Analysis 1: Comparison: Pregabalin; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

6. Primary Outcome: Change From Baseline in Daily Pain Score for NeP in PP Population at Week 6
Description: DPRS: participant rated 11-point Likert scale ranging from 0 (no pain) to 10 (worst possible pain) during past 24-hour period. Higher score indicates greater level of pain.
Time Frame: Baseline and Week 6
Population: PP population included participants who received the study medication for at least 6 weeks and indication of use was NeP.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 3087
Units on a scale
  Baseline | 5.58 (1.76)
  Change at Week 6 | -3.02 (1.75)
Statistical Analysis 1: Comparison: Pregabalin; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

7. Primary Outcome: Change From Baseline in Daily Pain Score for Fibromyalgia in ITT Population at Week 6
Description: as for outcome 6
Time Frame: Baseline and Week 6
Population: ITT population included participants who received at least 1 dose of the study medication and indication of use was fibromyalgia.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 120
Units on a scale
  Baseline | 6.69 (1.68)
  Change at Week 6 | -3.37 (1.74)
Statistical Analysis 1: Comparison: Pregabalin; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

8. Primary Outcome: Change From Baseline in Daily Pain Score for Fibromyalgia in PP Population at Week 6
Description: as for outcome 6
Time Frame: Baseline and Week 6
Population: PP population included participants who received the study medication for at least 6 weeks and indication of use was fibromyalgia.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 117
Units on a scale
  Baseline | 6.69 (1.69)
  Change at Week 6 | -3.37 (1.73)
Statistical Analysis 1: Comparison: Pregabalin; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

9. Secondary Outcome: Change From Baseline in Sleep Interference Score for NeP in ITT Population at Week 6
Description: Daily Sleep Interference Score (DSIS): participant rated 11-point Likert scale ranging from 0 (pain does not interfere with sleep) to 10 (pain completely interferes with sleep) during past 24-hour period. Higher score indicates a greater level of sleep disturbance. Self-assessment performed daily on awakening prior to taking study medication.
Time Frame: Baseline and Week 6
Population: ITT population included participants who received at least 1 dose of the study medication and indication of use was NeP.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 3210
Units on a scale
  Baseline | 4.25 (2.23)
  Change at Week 6 | -2.38 (1.89)
Statistical Analysis 1: Comparison: Pregabalin; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

10. Secondary Outcome: Change From Baseline in Sleep Interference Score for NeP in PP Population at Week 6
Description: DSIS: participant rated 11-point Likert scale ranging from 0 (pain does not interfere with sleep) to 10 (pain completely interferes with sleep) during past 24-hour period. Higher score indicates a greater level of sleep disturbance. Self-assessment performed daily on awakening prior to taking study medication.
Time Frame: Baseline and Week 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 3087
Units on a scale
  Baseline | 4.23 (2.22)
  Change at Week 6 | -2.37 (1.86)
Statistical Analysis 1: Comparison: Pregabalin; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

11. Secondary Outcome: Change From Baseline in Sleep Interference Score for Fibromyalgia in ITT Population at Week 6
Description: as for outcome 10
Time Frame: Baseline and Week 6
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 120
Units on a scale
  Baseline | 6.43 (1.80)
  Change at Week 6 | -3.19 (1.88)
Statistical Analysis 1: Comparison: Pregabalin; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

12. Secondary Outcome: Change From Baseline in Sleep Interference Score for Fibromyalgia in PP Population at Week 6
Description: as for outcome 10
Time Frame: Baseline and Week 6
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 117
Units on a scale
  Baseline | 6.41 (1.81)
  Change at Week 6 | -3.24 (1.82)
Statistical Analysis 1: Comparison: Pregabalin; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

13. Secondary Outcome: Number of Participants With Clinician's Global Impression of Change (CGIC) Scale for NeP in ITT Population
Description: CGIC: 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Change is defined as a score of 1 (very much improved), 2 (much improved), 3 (a little improved), 4 (no change), 5 (a little worse), 6 (much worse) or 7 (very much worse) on the scale. Higher score is equal to more affected.
Time Frame: Week 6
Population: ITT population included participants who received at least 1 dose of the study medication and indication of use was NeP.
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 3210
Participants
  Very much improved | 968
  Much improved | 1313
  A little improved | 671
  No change | 141
  A little worse | 7
  Much worse | 5
  Very much worse | 0

14. Secondary Outcome: Number of Participants With CGIC Scale for NeP in PP Population
Description: as for outcome 13
Time Frame: Week 6
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 3087
Participants
  Very much improved | 956
  Much Improved | 1306
  A little improved | 664
  No change | 140
  A little worse | 7
  Much worse | 5
  Very much worse | 0

15. Secondary Outcome: Number of Participants With Patient's Global Impression of Change (PGIC) Scale for NeP in ITT Population
Description: PGIC was defined as participant rated instrument to measure participant's change in overall status on a 7-point scale; range from 1 (very much improved) to 7 (very much worse). Change was defined as a score of 1 (very much improved), 2 (much improved), 3 (a little improved), 4 (no change), 5 (a little worse) , 6 (much worse) or 7 (very much worse) on the scale. Higher score is equal to more affected.
Time Frame: Week 6
Population: ITT population included participants who received at least 1 dose of the study medication and indication of use was NeP.
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 3210
Participants
  Very much improved | 1027
  Much improved | 1187
  A little improved | 686
  No change | 195
  A little worse | 5
  Much worse | 3
  Very much worse | 0

16. Secondary Outcome: Number of Participants With PGIC Scale for NeP in PP Population
Description: as for outcome 15
Time Frame: Week 6
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 3087
Participants
  Very much improved | 1018
  Much Improved | 1177
  A little improved | 680
  No change | 193
  A little worse | 5
  Much worse | 3
  Very much worse | 0

17. Secondary Outcome: Number of Participants With CGIC Scale for Fibromyalgia in ITT Population
Description: CGIC: 7-point clinician rated scale ranging from 1 (very much improved) to 7 (very much worse). Change was defined as a score of 1 (very much improved), 2 (much improved), 3 (a little improved), 4 (no change), 5 (a little worse), 6 (much worse) or 7 (very much worse) on the scale. Higher score is equal to more affected.
Time Frame: Week 6
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 120
Participants
  Very much improved | 30
  Much improved | 62
  A little improved | 21
  No change | 5
  A little worse | 0
  Much worse | 0
  Very much worse | 0

18. Secondary Outcome: Number of Participants With CGIC Scale for Fibromyalgia in PP Population
Description: as for outcome 17
Time Frame: Week 6
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 117
Participants
  Very much improved | 29
  Much Improved | 62
  A little improved | 21
  No change | 5
  A little worse | 0
  Much worse | 0
  Very much worse | 0

19. Secondary Outcome: Number of Participants With PGIC Scale for Fibromyalgia in ITT Population
Description: PGIC was defined as participant rated instrument to measure participant's change in overall status on a 7-point scale; range from 1 (very much improved) to 7 (very much worse). Change is defined as a score of 1 (very much improved), 2 (much improved), 3 (a little improved), 4 (no change), 5 (a little worse) , 6 (much worse) or 7 (very much worse) on the scale. Higher score is equal to more affected.
Time Frame: Week 6
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 120
Participants
  Very much improved | 35
  Much improved | 61
  A little improved | 14
  No change | 8
  A little worse | 0
  Much worse | 0
  Very much worse | 0

20. Secondary Outcome: Number of Participants With PGIC Scale for Fibromyalgia in PP Population
Description: as for outcome 19
Time Frame: Week 6
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 117
Participants
  Very much improved | 34
  Much Improved | 61
  A little improved | 14
  No change | 8
  A little worse | 0
  Much worse | 0
  Very much worse | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin
Serious Adverse Events (participants affected / at risk) | 2/4174
Other Adverse Events (participants affected / at risk) | 190/4174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=4174)
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=4174)
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 7
Diplopia (Eye disorders) | 2
Vision blurred (Eye disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 21
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Asthenia (General disorders) | 2
Chest pain (General disorders) | 2
Face oedema (General disorders) | 3
Fatigue (General disorders) | 3
Gait disturbance (General disorders) | 1
Oedema (General disorders) | 13
Oedema peripheral (General disorders) | 5
Pulmonary tuberculosis (Infections and infestations) | 2
Blood creatinine increased (Investigations) | 1
Blood glucose decreased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Weight increased (Investigations) | 1
Gout (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Increased appetite (Metabolism and nutrition disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 2
Cerebral infarction (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 4
Disturbance in attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 74
Headache (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 69
Speech disorder (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 1
Libido decreased (Psychiatric disorders) | 2
Sleep disorder (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 2
Skin disorder (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
It is highly likely that Adverse Events were under reported for this study as it was a Non Interventional study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.